CLINICAL TRIAL: NCT06052761
Title: Hospitalized Child and Play: Toys Made of Medical Materials
Brief Title: Child in Hospital and Playing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Maksude YILDIRIM, Research Assistant, Adiyaman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HRÜ/23.13.05
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Child in Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Making Toys from Medical Materials (Experimental): The purpose of the study will be explained to the children and their parents before the procedure, and verbal and written consent will be obtained from the parents who agree to participate in the study. Children's anxiety will be evaluated using the "Children's State Anxiety Scale (CSA)" before and after the procedure (half an hour after the first measurement), based on the statements of both the mother and the child.
  Interventions: Device: Making Toys from Medical Materials
- Control group (No Intervention): The purpose of the study will be explained to the children and their parents before the procedure, and verbal and written consent will be obtained from the parents who agree to participate in the study. No procedures will be performed other than routine procedures performed in the hospital. Children's anxiety will be evaluated based on the statements of both the mother and the child, using the "Children's State Anxiety Scale (CSA)" after obtaining consent from the parents and half an hour after the first measurement.

INTERVENTIONS:
Device: Making Toys from Medical Materials — Rabbit Making: The two fingers and the palm of the medical glove will be filled with cotton and the bottom part will be tied. The finger part of the glove will form the rabbit's ears, and the palm part will form its face. After the glove is shaped, the rabbit's eyes and mouth will be drawn with a pencil.
  Cat Making: Three abeslangs will be cut to appropriate sizes to create the cat. The cut pieces will be combined to form the cat's head, feet, and tail. After the assembly process is completed, the cat's eyes, nose and beard will be drawn with a pencil.
  Plane Making: The 10 cc syringe and needle tip removed from its packaging will be combined. Children will be asked to color the two abeslangs given to them in the color they want. The abeslangs painted by the children will be fixed to the syringe with a plaster, one on the bottom and the other on the top.
  Arms: Making Toys from Medical Materials

SUMMARY:
Being hospitalized is a stressful process for the child and her family. Management of stress is important to accelerate the child's recovery process and ensure early discharge. It is thought that playing with toys made using medical materials will reduce children's stress. This project aims to determine the effect of playing with toys made with medical materials on the stress of a hospitalized child. It is planned to collect the data of the project from pediatric patients aged 4-6 years hospitalized in the pediatric clinic of a training and research hospital in the Southeastern Anatolia Region. It is planned to analyze the data obtained from pediatric patients by using the SPSS program. As a result of the project, it is aimed that the game played with toys made using medical materials will reduce the stress of children.

DETAILED DESCRIPTION:
Children whose immune systems are not yet fully mature may encounter many acute or chronic diseases throughout their development and therefore may need to be hospitalized. Staying in an unknown environment such as a hospital causes children to experience feelings such as anxiety and fear.

Hospitalization, which is a stressful process for both the child and his family, causes financial and social changes for the child and his family. Being unfamiliar with the disease, the hospital environment, the procedures to be performed, and the feeling of not having control over the procedures also create stress on the child and the family. In addition to the stress experienced, the effects of their treatments on the central nervous system and the biological stress they bring negatively affect the development of hospitalized children. Hospitalized children experience different emotions due to the unknown environment, unfamiliar people in this environment, unknown tools and equipment, and frightening sounds and smells. For children, being sick and being hospitalized can easily lead to a crisis.

It is an indisputable fact that regardless of the age of the child, being separated from his family and hospitalized creates great stress for him. Effectively managing the stress of hospitalized children will shorten the hospitalization process by facilitating the child's adaptation to the disease and the hospital. When it comes to children, the first thing that comes to mind is play. For this reason, it is thought that the child will best cope with stress through play. It seems that play is an effective tool in helping hospitalized children cope with stress. When the literature was examined, studies were found examining the effects of games such as tablet games, outdoor games, and digital games on hospitalized children. In a study, the effect of playing with toys made with medical materials on the pain of children with cancer was evaluated. However, no study has been found examining the effect of playing with toys made using medical materials on the anxiety of hospitalized children. This study was planned as a randomized controlled study to examine the effect of playing with toys made of medical materials on the anxiety of hospitalized children.

ELIGIBILITY:
Inclusion Criteria:

* Children who are between the ages of 4-6,
* have no pain,
* have been hospitalized for at least two days,
* are receiving IV treatment, and
* whose parents approve of participating in the study will be included in the study.

Exclusion Criteria:

* Children with mental retardation who underwent surgical procedures will not be included in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Children's State Anxiety Scale (CSA) | 4 months
  This scale was developed in 2013 to measure the state anxiety of children in the 4-10 age group. The Turkish validity and reliability study of the scale was conducted in 2017. The scale is designed as a thermometer with a light bulb at the bottom and evenly spaced horizontal lines going up. Each horizontal line on the thermometer represents one point, and the bulb treasure at the bottom is 0 points. As you move up, the score obtained from the scale increases, and a maximum of 10 points is obtained. A score of 0 on the scale indicates no anxiety and a score of 10 indicates the highest anxiety. The scale can be used by creating different scenarios for children who understand the thermometer analogy and those who do not.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Faculty of Health Sciences, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I will decide after we start collecting study data.